CLINICAL TRIAL: NCT01365052
Title: A Multicenter, Randomized, Double-Blind, Placebo Controlled, Parallel Group Safety and Tolerability Trial of Naproxen Sodium/ Diphenhydramine Combination in an OTC Population
Brief Title: Safety Trial of Naproxen Sodium/ Diphenhydramine
Acronym: MUST
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple
Other Study IDs: 15560
Record Dates: First submitted 2011-05-17; First posted 2011-06-03 (Estimated); Results first posted 2014-06-16 (Estimated); Last update posted 2015-06-08 (Estimated); Status verified 2015-05

CONDITIONS: Pain
Keywords: Maximum Use Safety Trial
MeSH Terms: conditions — Pain | interventions — Naproxen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Naproxen sodium 440 mg/DPH 50 mg (BAY98-7111) (Experimental)
  Interventions: Drug: Naproxen sodium 440 mg/DPH 50 mg (BAY98-7111)
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Naproxen sodium 440 mg/DPH 50 mg (BAY98-7111) — 2 capsules each containing naproxen sodium 220 mg /diphenhydramine hydrochloride (DPH) 25 mg are taken orally with a full glass of water approximately 30 minutes prior to bedtime for 10 consecutive days
  Arms: Naproxen sodium 440 mg/DPH 50 mg (BAY98-7111)
Drug: Placebo — 2 placebo capsules are taken orally with a full glass of water 30 minutes prior to bedtime for 10 consecutive days
  Arms: Placebo

SUMMARY:
The purpose of this trial is to see how safe the combination of naproxen sodium 440 mg and diphenhydramine hydrochloride (DPH) 50 mg (the investigational product) is compared to placebo (capsules containing no drug) when taken for 10 days.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, ambulatory, male and female volunteers ages 12 and older
* History of experiencing occasional sleeplessness accompanied by aches and pains at least two times, but not continually for more than 14 days per month, in at least 2 of the past 3 months
* Female subjects of childbearing potential must be using a medically acceptable form of birth control, e.g., oral or patch contraceptives, intrauterine device, Depo-Provera®, for at least 1 month prior to screening (3 months on oral contraceptives), or double-barrier and have a negative pregnancy test at Screening. Female subjects of nonchildbearing potential must be amenorrheic for at least 2 years or have had a hysterectomy and/or bilateral oophorectomy
* Be willing and able to participate in all scheduled visits, treatment plan, tests and other trial procedures according to the protocol
* Provide a personally signed and dated informed consent indicating that the subject has been informed of all pertinent aspects of the trial, (subjects <18 years of age must sign a written assent and have parental or guardian consent).

Exclusion Criteria:

* History of hypersensitivity to naproxen sodium, acetaminophen, or any NSAIDs (Nonsteroidal Antiinflammatory Drugs), diphenhydramine or any other antihistamines, and similar pharmacological agents or components of the product
* Evidence or history of clinically significant (in the judgment of the investigator) hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic diseases, or malignancies with the last 5 years
* A history of a chronic or severe sleep problem which does not respond to OTC (Over-the-counter) medication and/or requires a prescription hypnotic or sedative
* Currently experiencing chronic pain or on chronic NSAID therapy (defined as taking a daily [5 to 7 days per week] regimen of prescription or OTC NSAIDs)
* Current or past history of gastrointestinal ulcers or bleeding or other bleeding disorders
* Use of any OTC or prescription medications with which the administration of naproxen, acetaminophen, or any NSAIDs, diphenhydramine or any other antihistamines or sedatives, is contraindicated
* Chronic use of other products containing diphenhydramine, including topical products
* Use of steroids or blood thinning (anticoagulant) drugs (aspirin 81 mg is permitted if the dose has been taken for at least one month prior to screening)

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 326 (Actual)
Dates: Start 2011-05; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (19):
- United States (19):
  - Chandler, Arizona
  - Mesa, Arizona
  - Peoria, Arizona
  - Anaheim, California
  - Rancho Cucamonga, California
  - Sacramento, California
  - Colorado Springs, Colorado
  - Kissimmee, Florida
  - Pembroke Pines, Florida
  - South Miami, Florida
  - Stockbridge, Georgia
  - Metairie, Louisiana
  - Elkridge, Maryland
  - Warwick, Rhode Island
  - Mt. Pleasant, South Carolina
  - Fort Worth, Texas
  - San Angelo, Texas
  - San Antonio, Texas
  - Salt Lake City, Utah

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Naproxen Sodium 440 mg/DPH 50 mg (BAY98-7111) | Placebo
Started | 217 | 109
Completed | 213 | 105
Not Completed | 4 | 4
Not completed — Adverse Event | 4 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Naproxen Sodium 440 mg/DPH 50 mg (BAY98-7111) | Placebo | Total
Number analyzed (Participants) | 217 | 109 | 326
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.9 (18.14) | 47.1 (19.26) | 47.0 (18.49)
Age, Customized [Number; unit: Participants] — Some categories will have overlapping samples
  Participants
    <60 years | 152 (70.0) | 72 (66.1) | 224
    Greater than or equal to 60 years | 65 (30.0) | 37 (33.9) | 102
    >65 years | 46 (21.2) | 28 (25.7) | 74
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 133 | 65 | 198
  Male | 84 | 44 | 128

OUTCOME MEASURES:

1. Other Pre Specified Outcome: Percentage of Subjects Who Discontinued Due to an Adverse Event for Those Subjects Who Are Randomized and Take at Least One Dose of Investigational Product
Time Frame: 10 days after randomization
Population: Safety population
Measure: Number; unit: Percentage of participants
Arm/Group | Naproxen Sodium 440 mg/DPH 50 mg (BAY98-7111) | Placebo
Number analyzed (Participants) | 217 | 109
Percentage of participants | 1.8 | 3.7

2. Primary Outcome: Percentage of Subjects With Any Adverse Event for Those Subjects Who Were Randomized and Took at Least One Dose of Investigational Product
Description: Please see further details in Adverse Events (AE) section
Time Frame: 10 days after randomization
Population: Safety population
Measure: Number; unit: Percentage of participants
Arm/Group | Naproxen Sodium 440 mg/DPH 50 mg (BAY98-7111) | Placebo
Number analyzed (Participants) | 217 | 109
Percentage of participants | 39.6 | 45.0

3. Primary Outcome: Percentage of Subjects With Any Serious Adverse Event for Those Subjects Who Were Randomized and Took at Least One Dose of Investigational Product
Description: Please see further details in AE section
Time Frame: 10 days after randomization
Population: Safety population
Measure: Number; unit: Percentage of participants
Arm/Group | Naproxen Sodium 440 mg/DPH 50 mg (BAY98-7111) | Placebo
Number analyzed (Participants) | 217 | 109
Percentage of participants | 0 | 0

4. Other Pre Specified Outcome: Treatment Compliance - Number of Capsules Taken
Time Frame: 10 days after randomization
Population: Safety population
Measure: Mean (Standard Deviation); unit: Capsules
Arm/Group | Naproxen Sodium 440 mg/DPH 50 mg (BAY98-7111) | Placebo
Number analyzed (Participants) | 217 | 109
Capsules | 20.1 (1.73) | 19.9 (2.98)

5. Other Pre Specified Outcome: Treatment Compliance - Duration of Exposure to Treatment in Days
Time Frame: 10 days after randomization
Population: Safety population
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Naproxen Sodium 440 mg/DPH 50 mg (BAY98-7111) | Placebo
Number analyzed (Participants) | 217 | 109
Days | 9.9 (0.76) | 9.8 (1.37)

ADVERSE EVENTS:
Time Frame: Treatment emergent adverse events (TEAEs) were collected from the date of the first dose of study drug in the treatment period for 12 days, or for 30 days after the last study drug administration if they were serious adverse events (SAEs).
Groups:
- Placebo: 2 over-encapsulated tablets of placebo are taken orally with a full glass of water 30 minutes prior to bedtime for 10 consecutive days
Arm/Group | Naproxen Sodium 440 mg/DPH 50 mg (BAY98-7111) | Placebo
Serious Adverse Events (participants affected / at risk) | 0/217 | 0/109
Other Adverse Events (participants affected / at risk) | 86/217 | 49/109
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Naproxen Sodium 440 mg/DPH 50 mg (BAY98-7111) (N=217) | Placebo (N=109)
ANISOCYTOSIS (Blood and lymphatic system disorders) | 0 | 1
HYPOCHROMASIA (Blood and lymphatic system disorders) | 0 | 1
MICROCYTOSIS (Blood and lymphatic system disorders) | 0 | 1
ANGINA PECTORIS (Cardiac disorders) | 0 | 1
EYE SWELLING (Eye disorders) | 1 | 0
VISION BLURRED (Eye disorders) | 1 | 0
ABDOMINAL DISCOMFORT (Gastrointestinal disorders) | 5 | 2
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 3 | 3
CONSTIPATION (Gastrointestinal disorders) | 1 | 1
DIARRHOEA (Gastrointestinal disorders) | 7 | 2
DRY MOUTH (Gastrointestinal disorders) | 1 | 1
DYSPEPSIA (Gastrointestinal disorders) | 5 | 1
DYSPHAGIA (Gastrointestinal disorders) | 1 | 0
FAECES DISCOLOURED (Gastrointestinal disorders) | 1 | 0
FLATULENCE (Gastrointestinal disorders) | 1 | 0
FREQUENT BOWEL MOVEMENTS (Gastrointestinal disorders) | 1 | 0
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 1 | 0
NAUSEA (Gastrointestinal disorders) | 9 | 1
OESOPHAGEAL DISCOMFORT (Gastrointestinal disorders) | 1 | 0
OESOPHAGEAL OEDEMA (Gastrointestinal disorders) | 1 | 0
OESOPHAGEAL PAIN (Gastrointestinal disorders) | 1 | 0
TOOTH LOSS (Gastrointestinal disorders) | 1 | 0
TOOTHACHE (Gastrointestinal disorders) | 3 | 2
VOMITING (Gastrointestinal disorders) | 1 | 0
ASTHENIA (General disorders) | 2 | 1
EARLY SATIETY (General disorders) | 1 | 0
FATIGUE (General disorders) | 2 | 0
OEDEMA PERIPHERAL (General disorders) | 1 | 0
PAIN (General disorders) | 2 | 1
PYREXIA (General disorders) | 1 | 0
SWELLING (General disorders) | 1 | 0
THIRST (General disorders) | 2 | 0
HYPERSENSITIVITY (Immune system disorders) | 1 | 0
SEASONAL ALLERGY (Immune system disorders) | 1 | 0
NASOPHARYNGITIS (Infections and infestations) | 0 | 1
PHARYNGITIS STREPTOCOCCAL (Infections and infestations) | 1 | 0
RHINITIS (Infections and infestations) | 1 | 0
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 | 0
URINARY TRACT INFECTION (Infections and infestations) | 2 | 1
VULVOVAGINAL MYCOTIC INFECTION (Infections and infestations) | 0 | 1
CONTUSION (Injury, poisoning and procedural complications) | 1 | 0
EXCORIATION (Injury, poisoning and procedural complications) | 1 | 0
LACERATION (Injury, poisoning and procedural complications) | 1 | 0
MUSCLE STRAIN (Injury, poisoning and procedural complications) | 1 | 1
ALANINE AMINOTRANSFERASE ABNORMAL (Investigations) | 1 | 0
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 1 | 0
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 1 | 0
BASOPHIL COUNT INCREASED (Investigations) | 0 | 1
BLOOD CREATININE INCREASED (Investigations) | 1 | 0
BLOOD GLUCOSE INCREASED (Investigations) | 1 | 0
BLOOD POTASSIUM INCREASED (Investigations) | 2 | 0
BLOOD UREA INCREASED (Investigations) | 1 | 0
BLOOD URINE PRESENT (Investigations) | 2 | 1
HAEMATOCRIT DECREASED (Investigations) | 0 | 1
HAEMOGLOBIN DECREASED (Investigations) | 0 | 1
HEART RATE INCREASED (Investigations) | 1 | 0
LYMPHOCYTE COUNT INCREASED (Investigations) | 0 | 1
NEUTROPHIL COUNT INCREASED (Investigations) | 0 | 1
RED BLOOD CELL COUNT INCREASED (Investigations) | 0 | 1
RED BLOOD CELLS URINE (Investigations) | 1 | 0
URINARY SEDIMENT PRESENT (Investigations) | 1 | 2
WEIGHT INCREASED (Investigations) | 1 | 0
WHITE BLOOD CELL COUNT INCREASED (Investigations) | 1 | 1
WHITE BLOOD CELLS URINE (Investigations) | 1 | 0
DECREASED APPETITE (Metabolism and nutrition disorders) | 1 | 0
FLUID RETENTION (Metabolism and nutrition disorders) | 0 | 1
GOUT (Metabolism and nutrition disorders) | 1 | 1
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 2 | 1
HYPERKALAEMIA (Metabolism and nutrition disorders) | 1 | 0
TYPE 2 DIABETES MELLITUS (Metabolism and nutrition disorders) | 0 | 1
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 1 | 1
BACK PAIN (Musculoskeletal and connective tissue disorders) | 8 | 3
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 0 | 1
MUSCLE TIGHTNESS (Musculoskeletal and connective tissue disorders) | 1 | 0
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 1 | 1
MUSCULOSKELETAL STIFFNESS (Musculoskeletal and connective tissue disorders) | 1 | 0
MYALGIA (Musculoskeletal and connective tissue disorders) | 2 | 0
NECK PAIN (Musculoskeletal and connective tissue disorders) | 2 | 0
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 | 0
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 0 | 4
DIZZINESS (Nervous system disorders) | 9 | 0
DYSGEUSIA (Nervous system disorders) | 1 | 0
HEADACHE (Nervous system disorders) | 23 | 21
HYPOAESTHESIA (Nervous system disorders) | 1 | 1
LETHARGY (Nervous system disorders) | 1 | 1
PSYCHOMOTOR HYPERACTIVITY (Nervous system disorders) | 1 | 0
RESTLESS LEGS SYNDROME (Nervous system disorders) | 1 | 0
SINUS HEADACHE (Nervous system disorders) | 1 | 0
SOMNOLENCE (Nervous system disorders) | 10 | 4
ANXIETY (Psychiatric disorders) | 1 | 0
DEPRESSION (Psychiatric disorders) | 1 | 0
INSOMNIA (Psychiatric disorders) | 3 | 1
RESTLESSNESS (Psychiatric disorders) | 3 | 1
GLYCOSURIA (Renal and urinary disorders) | 1 | 0
HAEMATURIA (Renal and urinary disorders) | 1 | 1
PYURIA (Renal and urinary disorders) | 0 | 1
DYSMENORRHOEA (Reproductive system and breast disorders) | 1 | 0
DRY THROAT (Respiratory, thoracic and mediastinal disorders) | 1 | 0
DYSPHONIA (Respiratory, thoracic and mediastinal disorders) | 0 | 1
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 | 1
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 2 | 0
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 4 | 3
RHINORRHOEA (Respiratory, thoracic and mediastinal disorders) | 1 | 0
RHONCHI (Respiratory, thoracic and mediastinal disorders) | 0 | 1
SINUS CONGESTION (Respiratory, thoracic and mediastinal disorders) | 2 | 0
SNEEZING (Respiratory, thoracic and mediastinal disorders) | 3 | 0
UPPER-AIRWAY COUGH SYNDROME (Respiratory, thoracic and mediastinal disorders) | 0 | 1
RASH (Skin and subcutaneous tissue disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days